CLINICAL TRIAL: NCT03999749
Title: A Phase II Study of the Interleukin-6 Receptor Inhibitor Tocilizumab in Combination With Ipilimumab and Nivolumab in Patients With Unresectable Stage III or Stage IV Melanoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-00008
Record Dates: First submitted 2019-06-25; First posted 2019-06-27 (Actual); Results first posted 2024-10-09 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Ipilimumab; Nivolumab; tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Induction Phase, Maintenance Phase (Experimental): Induction Phase: 2 induction treatment cycles of 42 days (6 weeks) each, of which the first cycle of 6 weeks is the dose-limiting toxicity (DLT) period.
  Maintenance Phase: Consists of treatment cycles of 84 days (12 weeks) each, and may extend up to 1 year.
  Interventions: Drug: Ipilimumab; Drug: Nivolumab; Drug: Tocilizumab

INTERVENTIONS:
Drug: Ipilimumab — 4 induction doses (during the 2 treatment cycles) at a dose of 1 mg/kg intravenously (IV) every 3 weeks, 4 times during the 12-week induction period, concurrent with nivolumab at 3 mg/kg administered at the same interval
Drug: Nivolumab — Nivolumab (3 mg/kg) will be administered IV on Days 1 and 22 of each 42-day induction treatment cycle. Nivolumab will continue to be administered IV at 240 mg flat dose every 2 weeks; i.e., at Days 1, 15, 29, 43, 57, and 71 of the 84-day treatment cycle for the first maintenance cycle until week 24, then nivolumab will be administered at 480 mg flat dose every 4 weeks to a maximum of 2 years
Drug: Tocilizumab — Administered intravenously for each 42-day induction treatment cycle. After 12 weeks of therapy, starting at Week 13, subjects enter the maintenance phase. Tocilizumab will be administered intravenously every 6 weeks during the first 84 day maintenance treatment cycle only at 4 mg/kg

SUMMARY:
This is a Phase II, open-label, single arm study. The study will consist of an assessment of the safety and tolerability of tocilizumab administered concurrently at 4 mg/kg every 6 weeks for 5 doses in combination with ipilimumab and nivolumab for four induction doses to week 12, then maintenance nivolumab alone up to one year to patients with advanced melanoma. Treatment will be divided into induction and maintenance phases. It is anticipated that this clinical study will inform the use of this 3-drug combination for further phase II and/or phase III clinical testing. The trial will include an assessment of the pharmacodynamic activity of tocilizumab administered in combination with ipilimumab and nivolumab.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have signed and dated an Institutional Review Board (IRB)/Independent Ethics Committee (IEC)-approved written informed consent form (ICF) in accordance with regulatory and institutional guidelines. This must be obtained before the performance of any protocol-related procedures that are not part of normal patient care.
* Patients must be willing and able to comply with scheduled visits, treatment schedule, laboratory tests, tumor biopsies, and other requirements of the study.
* All patients must be either Stage IIIb/c/d or Stage IV melanoma according to the American Joint Committee on Cancer (AJCC) (8th edition) and have histologically-confirmed melanoma that is felt to be surgically unresectable in order to be eligible. Please refer to the AJCC 8th edition Cancer Staging Manual for a description of tumor, lymph node, metastasis, and staging.
* All melanomas, except ocular/uveal melanoma, regardless of primary site of disease will be allowed; mucosal melanomas are eligible.
* Patients must not have received prior anticancer treatment for metastatic disease (for example, but not limited to, systemic, local, radiation, radiopharmaceutical).
* Exceptions: Surgery for melanoma and/or post-resection brain radiotherapy (RT) if Central Nervous System (CNS) metastases and adjuvant RT for locoregional disease after resection and/or prior treatment with adjuvant IFN-alpha, ipilimumab or nivolumab (as described in Exclusion Criterion 2).
* All patients must have their disease status documented by a complete physical examination and imaging studies within 4 weeks prior to the first dose of study drug. Imaging studies must include computerized tomography (CT) scan of chest, abdomen, pelvis, and all known sites of resected disease in the setting of Stage IIIb/c/d or Stage IV disease, and brain magnetic resonance imaging ([MRI]; brain CT is allowable if MRI is contraindicated).
* The complete set of baseline radiographic images must be available before treatment initiation.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
* Tumor tissue from the resected site of disease must be provided for biomarker analyses
* Prior treated CNS metastases must be without MRI evidence of recurrence for at least 4 weeks after treatment. Patients must be off immunosuppressive doses of systemic steroids (10 mg/day prednisone or equivalent) for at least 14 days prior to study drug administration, and must have returned to neurologic baseline status postoperatively.
* The 4-week period of stability is measured after the completion of the neurologic interventions (i.e., surgery and/or radiation).
* In addition to neurosurgery to treat CNS metastases, adjuvant radiation after the resection of CNS metastasis is allowed. Immunosuppressive doses of systemic steroids (doses > 10 mg/day prednisone or equivalent) must be discontinued at least 14 days before study drug administration.
* Prior surgery that required general anesthesia must be completed at least 4 weeks before study drug administration. Surgery requiring local/epidural anesthesia must be completed at least 72 hours before study drug administration.
* Normal labs
* Patient Re-enrollment: This study permits the re-enrollment of a patient that has discontinued the study as a screen failure (i.e., patient has not been dosed/has not been treated). If re-enrolled, the patient must be re-consented and satisfy all eligibility criteria.
* Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [human chorionic gonadotropin (hCG)] hormone) within 24 hours prior to the start of study drug.
* Women of childbearing potential must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug(s) plus 5 half-lives of study drug plus 30 days (duration of ovulatory cycle). The half-life of nivolumab and ipilimumab is up to 25 days and 18 days, respectively. WOCBP should therefore use an adequate method to avoid pregnancy for a total of 23 weeks post treatment completion (Section 4.5).
* Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug(s) plus 5 half lives of the study drug (s) plus 90 days (duration of sperm turnover). The half lives of nivolumab and ipilimumab are up to 25 days and 18 days, respectively. Men should therefore use an adequate method of contraception for a total of 31 weeks post treatment completion (Section 4.5).
* Azoospermic males and WOCBP who are continuously not heterosexually active are exempt from contraceptive requirements. However, they must still undergo pregnancy testing as described in this section.

Exclusion Criteria:

* Patients with carcinomatosis meningitis or a history of current ocular/uveal melanoma are excluded.
* Patients with previous nonmelanoma malignancies are excluded unless a complete resection or remission was achieved at least 2 years prior to study entry and no additional therapy is required or anticipated to be required during the study period (exceptions include, but are not limited to, nonmelanoma skin cancers, in situ bladder cancer, in situ gastric cancer or gastrointestinal stromal tumor, in situ colon cancers, in situ cervical cancers/dysplasia, or breast carcinoma in situ).
* Patients with active, known, or suspected autoimmune disease. Patients with type I diabetes mellitus, residual hypothyroidism due to autoimmune thyroiditis only requiring hormone replacement, or skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment are permitted to enroll. For any cases of uncertainty, it is recommended that the Principal Investigator be consulted prior to signing informed consent.
* Patients with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone or equivalent) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids are permitted in the absence of active autoimmune disease.
* Prior therapy for melanoma with the following exceptions which are allowed: 1) surgery for the melanoma lesion(s), 2) adjuvant RT after neurosurgical resection for CNS lesions or for resected locoregional disease, and 3) prior adjuvant interferon (IFN)-alpha, ipilimumab and nivolumab (see qualifier below).
* Prior treatment with adjuvant IFN-alpha, adjuvant ipilimumab and/or nivolumab are allowed if completed 6 months prior to treatment.
* Treatment directed against the melanoma (eg, chemotherapy, targeted agents, biotherapy, limb perfusion) that is administered after a prior complete resection other than adjuvant radiation after neurosurgical resection or resection of locoregional disease and IFN-alpha, ipilimumab and nivolumab for resected melanoma.
* abnormalities labs
* Corrected QT interval using Fridericia's formula value > 480 msec at screening; family or personal history of long corrected QT interval (QTc) syndrome or ventricular arrhythmias including ventricular bigeminy at screening; previous history of drug induced QTc prolongation or the need for treatment with medications known or suspected of producing prolonged QTc intervals on electrocardiogram (ECG).
* Congestive heart failure (New York Heart Association Class III or IV), myocardial infarction
* Any serious or uncontrolled medical disorder or active infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2019-06-11 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2030-04-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Janice Mehnert, MD, Principal Investigator — New York Langone Health
Locations (4):
- United States (4):
  - The Angeles Clinic, Los Angeles, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - NYU Langone Health, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: janice.mehnert@nyulangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be provided access upon reasonable request. Requests should be directed to janice.mehnert@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Fa'ak F, Buni M, Falohun A, Lu H, Song J, Johnson DH, Zobniw CM, Trinh VA, Awiwi MO, Tahon NH, Elsayes KM, Ludford K, Montazari EJ, Chernis J, Dimitrova M, Sandigursky S, Sparks JA, Abu-Shawer O, Rahma O, Thanarajasingam U, Zeman AM, Talukder R, Singh N, Chung SH, Grivas P, Daher M, Abudayyeh A, Osman I, Weber J, Tayar JH, Suarez-Almazor ME, Abdel-Wahab N, Diab A. Selective immune suppression using interleukin-6 receptor inhibitors for management of immune-related adverse events. J Immunother Cancer. 2023 Jun;11(6):e006814. doi: 10.1136/jitc-2023-006814. PMID 37328287

RESULTS

PARTICIPANT FLOW:
Groups:
- Induction Phase, Maintenance Phase: Induction Phase: 2 induction treatment cycles of 42 days (6 weeks) each, of which the first cycle of 6 weeks is the dose-limiting toxicity (DLT) period.
  Maintenance Phase: Consists of treatment cycles of 84 days (12 weeks) each, and may extend up to 1 year.
  Ipilimumab: 4 induction doses (during the 2 treatment cycles) at a dose of 1 mg/kg intravenously (IV) every 3 weeks, 4 times during the 12-week induction period, concurrent with nivolumab at 3 mg/kg administered at the same interval
  Nivolumab: Nivolumab (3 mg/kg) will be administered IV on Days 1 and 22 of each 42-day induction treatment cycle. Nivolumab will continue to be administered IV at 240 mg flat dose every 2 weeks; i.e., at Days 1, 15, 29, 43, 57, and 71 of the 84-day treatment cycle for the first maintenance cycle until week 24, then nivolumab will be administered at 480 mg flat dose every 4 weeks to a maximum of 2 years
  Tocilizumab: Administered intravenously for each 42-day induction treatment cycle. After 12 weeks of therapy, starting at Week 13, subjects enter the maintenance phase. Tocilizumab will be administered intravenously every 6 weeks during the first 84 day maintenance treatment cycle only at 4 mg/kg
Period: Overall Study
Arm/Group | Induction Phase, Maintenance Phase
Started | 71
Completed | 16
Not Completed | 55
Not completed — Toxicity | 16
Not completed — Withdrawal by Subject | 3
Not completed — Disease progression | 26
Not completed — Physician Decision | 4
Not completed — Death | 5
Not completed — Patient deemed ineligible after treatment | 1

BASELINE CHARACTERISTICS:
Groups:
- Induction Phase, Maintenance Phase: Induction Phase: 2 induction treatment cycles of 42 days (6 weeks) each, of which the first cycle of 6 weeks is the DLT period.
  Maintenance Phase: Consists of treatment cycles of 84 days (12 weeks) each, and may extend up to 1 year.
  Ipilimumab: 4 induction doses (during the 2 treatment cycles) at a dose of 1 mg/kg intravenously (IV) every 3 weeks, 4 times during the 12-week induction period, concurrent with nivolumab at 3 mg/kg administered at the same interval
  Nivolumab: Nivolumab (3 mg/kg) will be administered IV on Days 1 and 22 of each 42-day induction treatment cycle. Nivolumab will continue to be administered IV at 240 mg flat dose every 2 weeks; i.e., at Days 1, 15, 29, 43, 57, and 71 of the 84-day treatment cycle for the first maintenance cycle until week 24, then nivolumab will be administered at 480 mg flat dose every 4 weeks to a maximum of 2 years
  Tocilizumab: Administered intravenously for each 42-day induction treatment cycle. After 12 weeks of therapy, starting at Week 13, subjects enter the maintenance phase. Tocilizumab will be administered intravenously every 6 weeks during the first 84 day maintenance treatment cycle only at 4 mg/kg
Arm/Group | Induction Phase, Maintenance Phase
Number analyzed (Participants) | 16
Age, Continuous [Median (Standard Deviation); unit: years] | 64.5 (11.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 13
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Grades 3-5 Treatment Related Immune Related Adverse Events (irAEs)
Description: Adverse events are graded according to the NCI CTCAE version 5.0. Immune-related adverse events (irAEs) are specific events occurring within 100 days of the last dose (which includes pneumonitis, diarrhea/colitis, hepatitis, nephritis/renal dysfunction, rash, and endocrine abnormalities [adrenal insufficiency, hypothyroidism/thyroiditis, hyperthyroidism, diabetes mellitus, and hypophysitis]), regardless of causality, for which patients received immunosuppressive medication for treatment of the event. The exception to the immunosuppressive medication criteria for irAEs is endocrine events (e.g., hypothyroidism/thyroiditis, hyperthyroidism, hypophysitis, diabetes mellitus, adrenal insufficiency), which are included regardless of treatment since these events are often managed without immunosuppression.
Time Frame: From start of treatment up to 100 days post treatment, *up to 18 months*
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Induction Phase, Maintenance Phase
Number analyzed (Participants) | 70
percentage of participants | 22.9 [13.7 to 34.5]

2. Primary Outcome: Objective Response Rate (ORR)
Description: Objective Response Rate (ORR) is defined as the total number of patients whose best response outcome is a CR or PR by week 24 divided by the total number of evaluable patients. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Week 24
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Induction Phase, Maintenance Phase
Number analyzed (Participants) | 70
percentage of participants | 48.6 [36.5 to 60.9]

3. Secondary Outcome: Disease Control Rate (DCR)
Description: Disease Control Rate (DCR) is defined as the total number of patients whose best response outcome is a complete response (CR) or partial response (PR), or SD divided by the total number of evaluable patients.
Time Frame: From beginning of treatment until the first observation of disease progression (up to 5 years)
Reporting Status: Not Posted, anticipated posting 2031-04

4. Secondary Outcome: Progression-Free Survival (PFS)
Description: Progression-Free Survival (PFS) is defined for each patient as the time from first dosing to the first observation of disease progression or death due to any cause. If a patient has not progressed or died at the time of analysis, PFS will be censored on the date of the last disease assessment. Patients who do not have any tumor assessment on treatment will be censored on the day of the first dose.
Time Frame: From start of treatment until the first observation of disease progression or death due to any cause, whichever came first (up to 5 years)
Reporting Status: Not Posted, anticipated posting 2031-04

5. Secondary Outcome: Duration of Overall Response
Description: Duration of Overall Response will be computed for all patients whose best response is either a PR or CR and is calculated from the time the measurement criteria are met for PR or CR, whichever is recorded first, until the date of documented PD or death.
Time Frame: From date of best overall response until the first observation of disease progression or death due to any cause, whichever came first (up to 5 years)
Reporting Status: Not Posted, anticipated posting 2031-04

6. Secondary Outcome: Duration of Disease Control
Description: Duration of Disease Control will be computed for the patients who had ORR outcome of CR, PR, or SD and is calculated from the beginning of treatment until the time of documented disease progression.
Time Frame: From start of treatment until the first observation of disease progression (up to 5 years)
Reporting Status: Not Posted, anticipated posting 2031-04

7. Secondary Outcome: Immune-related Response Rate (irRR)
Description: Immune-related Response Rate (irRR) is defined as the proportion of response evaluable patients whose Immune Related Best Overall Response (irBOR) outcome is irPR, irCR.
Time Frame: From beginning of treatment until the first observation of disease progression (up to 5 years)
Reporting Status: Not Posted, anticipated posting 2031-04

8. Secondary Outcome: Immune-related Disease Control Rate
Description: Immune-related Disease Control Rate is defined as the proportion of the response evaluable patients whose irBOR outcome is irPR, irCR, or immune-related stable disease (irSD).
Time Frame: From beginning of treatment until the first observation of disease progression (up to 5 years)
Reporting Status: Not Posted, anticipated posting 2031-04

9. Secondary Outcome: Immune-related Progression-Free Survival (irPFS)
Description: Immune-related Progression-Free Survival (irPFS) is defined as the time between the first dosing date and the date of immune-related progressive disease (irPD) or death, whichever occurs first. For patients with no recorded post-baseline tumor assessment, irPFS will be censored at the day of first dose. A patient who dies without reported irPD will be considered to have progressed on the date of death. For those who remain alive and have no irPD, irPFS will be censored on the date of last evaluable tumor assessment. Patients who do not have any tumor assessment on treatment will be censored on the day of the first dose.
Time Frame: as for outcome 4
Reporting Status: Not Posted, anticipated posting 2031-04

10. Secondary Outcome: Duration of Immune-related Overall Response
Description: Duration of Immune-related Overall Response will be computed for all patients whose irBOR outcome is either an irPR or irCR and is calculated from the time the measurement criteria are met for irPR or irCR, whichever is recorded first, until the date of documented PD or death by irRC.
Time Frame: From time irPR or irCR was met until the first observation of disease progression or death due to any cause, whichever came first (up to 5 years)
Reporting Status: Not Posted, anticipated posting 2031-04

11. Secondary Outcome: Duration of Immune-related Disease Control
Description: Duration of Immune-related Disease Control will be computed for the patients who had irBOR outcome of irCR, irPR, or irSD and is calculated from the beginning of treatment until the time of documented disease progression by irRC.
Time Frame: From beginning of treatment until the first observation of disease progression (up to 5 years)
Reporting Status: Not Posted, anticipated posting 2031-04

12. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival is defined for each patient as the time from first dosing to death due to any cause. If a patient has not died at the time of analysis, OS will be censored as of their last known date alive (i.e. last time patient was contacted for any reason in the study). Patients who do not have any tumor assessment on treatment be followed up for OS, and their date of death will be incorporated into the OS analysis.
Time Frame: From start of treatment until the date of death from any cause (up to 5 years)
Reporting Status: Not Posted, anticipated posting 2031-04

ADVERSE EVENTS:
Time Frame: AEs are assessed up to 59 weeks. SAEs are assessed up to 18 months. All-Cause Mortality is assessed up to 5 years.
Description: PI monitors for AEs at every follow-up visit
Arm/Group | Induction Phase, Maintenance Phase
All-Cause Mortality (participants affected / at risk) | 22/71
Serious Adverse Events (participants affected / at risk) | 34/71
Other Adverse Events (participants affected / at risk) | 71/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Induction Phase, Maintenance Phase (N=71)
Anemia (Blood and lymphatic system disorders) | 4
Lymphopenia (Blood and lymphatic system disorders) | 1
Bradycardia (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Adrenal Insufficiency (Endocrine disorders) | 2
Dislocated Iris (Eye disorders) | 1
Infection (Eye disorders) | 1
Incarcerated Hernia (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 6
ABD pain (Gastrointestinal disorders) | 2
Colitis (Gastrointestinal disorders) | 2
Duodenal Hemorrhage (Gastrointestinal disorders) | 1
Anal Hemorrhage (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Enteritis (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Weakness (General disorders) | 1
Death (General disorders) | 2
Checkpoint inhibitor hepatitis (Hepatobiliary disorders) | 1
Immune Checkpoint Inhibitor Hepatitis (Hepatobiliary disorders) | 1
COVID-19 infection (Infections and infestations) | 1
COVID-19 Pneumonia (Infections and infestations) | 2
Lyme Disease (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
UTI (Infections and infestations) | 1
Lung Infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 3
Shingles (Infections and infestations) | 1
Skin Infection (Infections and infestations) | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1
ALT increase (Investigations) | 6
Alkaline phosphate increase (Investigations) | 1
AST increase (Investigations) | 5
Blood bilirubin increase (Investigations) | 1
Creatinine increase (Investigations) | 2
GGT increase (Investigations) | 2
Lipase increase (Investigations) | 6
Lymphocyte count increase (Investigations) | 1
Neutrophil count decreased (Investigations) | 2
Platelet count decrease (Investigations) | 1
Serum amylase increased (Investigations) | 2
Hypercalcemia (Metabolism and nutrition disorders) | 1
Acidosis (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 3
Hypermagnesemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 3
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 3
Generalized Muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Arthalgia (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 4
Stroke (Nervous system disorders) | 2
Confusion (Psychiatric disorders) | 1
Acute Kidney injury (Renal and urinary disorders) | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Adult respirartory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1
Diffuse dermatitis (Skin and subcutaneous tissue disorders) | 1
Incarcerated Hernia Repair (Surgical and medical procedures) | 1
Sinus Surgery with Septoplasty (Surgical and medical procedures) | 1
Hypotension (Vascular disorders) | 2
Thromboembolic event (Vascular disorders) | 2
Hot flashes (Vascular disorders) | 8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Induction Phase, Maintenance Phase (N=71)
Anemia (Blood and lymphatic system disorders) | 17
Lymph Node Pain (Blood and lymphatic system disorders) | 1
Eosinophilia (Blood and lymphatic system disorders) | 2
Transaminitis (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Hypovolemia (Blood and lymphatic system disorders) | 1
increased L inguinal Lesion pain (Blood and lymphatic system disorders) | 1
Platelet count decreased (Blood and lymphatic system disorders) | 1
Hypertension (Blood and lymphatic system disorders) | 1
Elevated Eosinophils (Blood and lymphatic system disorders) | 1
Ventricular dysfunction with left ventricular hypertrophy (Cardiac disorders) | 1
Reduced e' velocities on ECHO (Cardiac disorders) | 1
Ventricular arrhythmia (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 1
Palpatations (Cardiac disorders) | 3
Cyanosis (Cardiac disorders) | 1
Chest Pain (Cardiac disorders) | 4
Tinnitus (Ear and labyrinth disorders) | 1
Hearing impaired (Ear and labyrinth disorders) | 2
impacted cerumen (Ear and labyrinth disorders) | 1
Otitis (Ear and labyrinth disorders) | 1
Hearing loss (Ear and labyrinth disorders) | 1
Ear Pain (Ear and labyrinth disorders) | 3
Hypopituitarism (Endocrine disorders) | 1
Hypophysitis (Endocrine disorders) | 5
Testosterone deficiency (Endocrine disorders) | 3
Adrenal Insufficiency (Endocrine disorders) | 7
Hyperthyroidism (Endocrine disorders) | 8
Hypothyroidism (Endocrine disorders) | 11
Blurred vision (Eye disorders) | 5
Glaucoma (Eye disorders) | 1
Eye Pain (Eye disorders) | 1
Uveitis (Eye disorders) | 3
Watering eyes (Eye disorders) | 3
Cataracts (Eye disorders) | 1
Photophobia (Eye disorders) | 2
Dry eyes (Eye disorders) | 5
Floaters (Eye disorders) | 1
Broken Blood vessel (Eye disorders) | 1
Eye Itching (Eye disorders) | 1
Ocular Migraine (Eye disorders) | 1
R. Eye Stye (Eye disorders) | 1
Eye Irritation (Eye disorders) | 1
R. Eye Hordeolum (Eye disorders) | 1
Rectal Pain (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 31
Enterocolitis (Gastrointestinal disorders) | 2
Pancreatitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 14
Bloating (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 34
ABD pain (Gastrointestinal disorders) | 14
Vomiting (Gastrointestinal disorders) | 10
Dry mouth (Gastrointestinal disorders) | 7
Stomach Pain (Gastrointestinal disorders) | 2
Gastritis (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 4
Dysphagia (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 2
Mucositis oral (Gastrointestinal disorders) | 2
Oral Pain (Gastrointestinal disorders) | 3
Hematochezia (Gastrointestinal disorders) | 1
Tubular adenoma in colon (Gastrointestinal disorders) | 1
Thickened Ileum (Gastrointestinal disorders) | 1
Loose Stool (Gastrointestinal disorders) | 3
Soft Stool (Gastrointestinal disorders) | 1
Tooth Extraction (Gastrointestinal disorders) | 1
Mouth Ulcers (Gastrointestinal disorders) | 1
Left Upper Quadrant discomfort (Gastrointestinal disorders) | 1
Phlegm (Gastrointestinal disorders) | 1
Diverticulitis (Gastrointestinal disorders) | 1
Barrett's Esophagus (Gastrointestinal disorders) | 1
Motion sickness (Gastrointestinal disorders) | 1
Mouth sores (Gastrointestinal disorders) | 1
Early Satiety (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Edema Limbs (General disorders) | 16
Fatigue (General disorders) | 40
Fever (General disorders) | 12
Night Sweats (General disorders) | 1
Injection site reaction (General disorders) | 1
Edema face (General disorders) | 1
Pain (General disorders) | 17
Edema trunk (General disorders) | 1
Chills (General disorders) | 7
Malaise (General disorders) | 2
Non-cardiac chest pain (General disorders) | 3
R sided pain (General disorders) | 1
Localized edema (General disorders) | 3
Flu-like symptoms (General disorders) | 4
R Arm pain (General disorders) | 1
R Neck pain (General disorders) | 1
Groin Pain (General disorders) | 1
Groin Abscess (General disorders) | 1
Post-op pain (General disorders) | 1
R toe pain (General disorders) | 1
Leg pain (General disorders) | 1
Swelling (General disorders) | 1
Vaccination site lymphadenopathy (General disorders) | 1
Left hip pain (General disorders) | 1
Injection realated reaction (General disorders) | 1
COVID-19 (General disorders) | 1
Intermittent hemoptysis (General disorders) | 1
Weakness (General disorders) | 1
Transaminitis (Hepatobiliary disorders) | 1
Allergic reaction (Immune system disorders) | 1
Allergic reaction to contrast (Immune system disorders) | 1
Folliculitis (Infections and infestations) | 1
Herpes Simplex reactivation (Infections and infestations) | 1
Enterocolitis infectious (Infections and infestations) | 1
Conjunctivitis (Infections and infestations) | 1
Shingles (Infections and infestations) | 4
Otitis externa (Infections and infestations) | 1
Prostate infection (Infections and infestations) | 1
Otitis media (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Vulval infection (Infections and infestations) | 1
UTI (Infections and infestations) | 5
Upper Respiratory Infection (Infections and infestations) | 7
Tooth infection (Infections and infestations) | 2
Papulopustular rash (Infections and infestations) | 2
Skin Infection (Infections and infestations) | 4
COVID-19 (Infections and infestations) | 4
Diverticulitis (Infections and infestations) | 1
Fungal infection (Infections and infestations) | 1
GI Virus (Infections and infestations) | 1
Lower leg cellulitis (Infections and infestations) | 1
Left foot fungal infection (Infections and infestations) | 1
Tinea Pedis (Infections and infestations) | 1
Left Mycotic Nail (Infections and infestations) | 1
Lyme disease (Infections and infestations) | 1
Latent tuberculosis (Infections and infestations) | 1
Influenza A (Infections and infestations) | 1
Thrush (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 2
Infusion related reacton (Injury, poisoning and procedural complications) | 10
Seroma (Injury, poisoning and procedural complications) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Umbilical Hernia (Injury, poisoning and procedural complications) | 1
Pressure ulcers (Injury, poisoning and procedural complications) | 1
Left knee meniscus tear (Injury, poisoning and procedural complications) | 1
Dermatitis (Injury, poisoning and procedural complications) | 1
Insect Bite (Injury, poisoning and procedural complications) | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1
Steroid Withdrawal (Injury, poisoning and procedural complications) | 1
Activated partial thromboplastin prolonged (Investigations) | 1
ALT increase (Investigations) | 25
Alkaline phosphate increase (Investigations) | 10
AST increase (Investigations) | 28
Blood bilirubin increase (Investigations) | 4
LDH increase (Investigations) | 11
Cardiac troponin T increase (Investigations) | 3
Cholesterol high (Investigations) | 1
Creatinine increase (Investigations) | 12
GGT increase (Investigations) | 12
Lipase increase (Investigations) | 18
Lymphocyte count decrease (Investigations) | 1
Neutrophil count decreased (Investigations) | 9
Pancreatic enzymes decrease (Investigations) | 1
Platelet count decrease (Investigations) | 9
Serum Amylase increase (Investigations) | 18
Thyroid stimulating hormone increased (Infections and infestations) | 5
Weight gain (Investigations) | 1
Weight loss (Investigations) | 6
White blood cell count decrease (Investigations) | 6
Headaches (Investigations) | 1
Transaminitis (Investigations) | 2
Acidosis (Metabolism and nutrition disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 12
Decreased appetite (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 7
Hyperkalemia (Metabolism and nutrition disorders) | 8
Hyponatremia (Metabolism and nutrition disorders) | 15
Hypernatremia (Metabolism and nutrition disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 5
Hyperphosphatemia (Metabolism and nutrition disorders) | 9
Hypercalcemia (Metabolism and nutrition disorders) | 5
Hypermagnesemia (Metabolism and nutrition disorders) | 1
Hyperuricemia (Metabolism and nutrition disorders) | 6
Hypoalbuminemia (Metabolism and nutrition disorders) | 8
Hypocalcemia (Metabolism and nutrition disorders) | 4
Hypokalemia (Metabolism and nutrition disorders) | 9
Hypomagnesemia (Metabolism and nutrition disorders) | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 5
R. Knee Pain (Musculoskeletal and connective tissue disorders) | 1
Left side Rib Pain (Musculoskeletal and connective tissue disorders) | 1
Myoclonus (Musculoskeletal and connective tissue disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1
Trigger finger (Musculoskeletal and connective tissue disorders) | 2
Bursitis (Musculoskeletal and connective tissue disorders) | 2
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Pain from lung resection site (Musculoskeletal and connective tissue disorders) | 1
muscle cramp (Musculoskeletal and connective tissue disorders) | 4
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9
Myalgia (Musculoskeletal and connective tissue disorders) | 13
Arthalgia (Musculoskeletal and connective tissue disorders) | 22
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 8
Flank pain (Musculoskeletal and connective tissue disorders) | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 5
Groin Pain (Musculoskeletal and connective tissue disorders) | 1
Ovarian Cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Presumed Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Abnormal lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lumbar radiculopathy (Nervous system disorders) | 1
Post shingles neuropathy (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 16
Headache (Nervous system disorders) | 20
Peripheral motor neuropathy (Nervous system disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 6
Paresthesia (Nervous system disorders) | 6
Sciatica (Nervous system disorders) | 1
Concentration impairment (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 2
Neuralgia (Nervous system disorders) | 1
Lethargy (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 3
Stroke (Nervous system disorders) | 2
Syncope (Nervous system disorders) | 1
Lightheadedness (Nervous system disorders) | 1
Ulnar neuropathy (Nervous system disorders) | 1
Mood changes (Psychiatric disorders) | 1
Agitation (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 4
Insomnia (Psychiatric disorders) | 17
Anxiety (Psychiatric disorders) | 3
Confusion (Psychiatric disorders) | 2
Chronic kidney disease (Renal and urinary disorders) | 1
Renal colic (Renal and urinary disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Glucosuria (Renal and urinary disorders) | 1
Cystitis (Renal and urinary disorders) | 1
Urinary Retention (Renal and urinary disorders) | 2
Urinary Hesitancy (Renal and urinary disorders) | 1
Renal hesitancy (Renal and urinary disorders) | 1
Polyuria (Renal and urinary disorders) | 1
Urine Discoloration (Renal and urinary disorders) | 2
Urinary incontinence (Renal and urinary disorders) | 1
Urinary tract pain (Renal and urinary disorders) | 1
Urinary frequency (Renal and urinary disorders) | 2
Bilateral hydronephrosis (Renal and urinary disorders) | 1
Acute Kidney injury (Renal and urinary disorders) | 1
Vaginal dryness (Reproductive system and breast disorders) | 3
Pelvic pain (Reproductive system and breast disorders) | 1
Prostatomegaly (Reproductive system and breast disorders) | 1
Perineal soreness (Reproductive system and breast disorders) | 1
Erectile dysfunction (Reproductive system and breast disorders) | 2
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 5
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 3
Cough (Renal and urinary disorders) | 18
Breathing tightness (Respiratory, thoracic and mediastinal disorders) | 1
Flu-like symptom (Respiratory, thoracic and mediastinal disorders) | 1
Intermittent hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3
Pleaural Effusion (Respiratory, thoracic and mediastinal disorders) | 3
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 2
Rales (Respiratory, thoracic and mediastinal disorders) | 1
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 2
Post nasal drip (Respiratory, thoracic and mediastinal disorders) | 2
COVID-19 (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 12
Scalp abrasion (Skin and subcutaneous tissue disorders) | 1
Scalp lesion (Skin and subcutaneous tissue disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 3
Eczema Skin Roughness (Skin and subcutaneous tissue disorders) | 2
Lesions (axilla + breast) (Skin and subcutaneous tissue disorders) | 1
Erythematous rash (Skin and subcutaneous tissue disorders) | 2
Micronodular BCC (Skin and subcutaneous tissue disorders) | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 4
Lichenoid dermatitis (Skin and subcutaneous tissue disorders) | 1
Asteatotic dermatitis (Skin and subcutaneous tissue disorders) | 1
Subcutaneous nodule (Skin and subcutaneous tissue disorders) | 1
Pityriasis (Skin and subcutaneous tissue disorders) | 1
Purpura (Skin and subcutaneous tissue disorders) | 1
Tick bite (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 9
Alopecia (Skin and subcutaneous tissue disorders) | 2
Pain of skin (Skin and subcutaneous tissue disorders) | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2
Intertrigo groin (Skin and subcutaneous tissue disorders) | 1
Tinea corporis (Skin and subcutaneous tissue disorders) | 1
Tinea pedis (Skin and subcutaneous tissue disorders) | 2
Hives (Skin and subcutaneous tissue disorders) | 1
Redness (Skin and subcutaneous tissue disorders) | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 12
Pruritis (Skin and subcutaneous tissue disorders) | 36
Fungal rash (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 31
SCC left chest (Skin and subcutaneous tissue disorders) | 1
Eyelid skin tag (Skin and subcutaneous tissue disorders) | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 2
Inflamed keratosis (Skin and subcutaneous tissue disorders) | 1
Grover's disease (Skin and subcutaneous tissue disorders) | 1
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 1
Sehorrheic keratosis (Skin and subcutaneous tissue disorders) | 1
Diffuse dermatitis (Skin and subcutaneous tissue disorders) | 1
Left fore-arm nodule (Skin and subcutaneous tissue disorders) | 1
Lip nodule (Skin and subcutaneous tissue disorders) | 1
Rash from poison sumac (Skin and subcutaneous tissue disorders) | 1
Vitiligo (Skin and subcutaneous tissue disorders) | 1
SCC (Surgical and medical procedures) | 1
Lung Resection (Surgical and medical procedures) | 1
Cataract (Surgical and medical procedures) | 1
Root canal (Surgical and medical procedures) | 1
Endoscopic retrograde cholangiopancreatography (Surgical and medical procedures) | 1
Excision of ABD wall mass (Surgical and medical procedures) | 1
Flushing (Vascular disorders) | 1
Hypertension (Vascular disorders) | 2
Hypotension (Vascular disorders) | 2
Lymphedema (Vascular disorders) | 1
Right Lower Extremity DVT (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must review and approve any results of the study or abstracts for professional meetings prepared by the Investigator. Published data must not compromise the objectives of the study. Data from individual study centers in multicenter studies must not be published separately.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-13): https://cdn.clinicaltrials.gov/large-docs/49/NCT03999749/Prot_SAP_000.pdf